CLINICAL TRIAL: NCT03411681
Title: Resistance Exercise as a Strategy to Enhance Postprandial Muscle Protein Synthesis in Obese Adults
Brief Title: Resistance Exercise and Muscle Protein Synthesis in Obese Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16699
Record Dates: First submitted 2017-12-12; First posted 2018-01-26 (Actual); Last update posted 2018-05-01 (Actual); Status verified 2017-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Weight (Active Comparator)
  Interventions: Other: Resistance Exercise
- Obese (Experimental)
  Interventions: Other: Resistance Exercise

INTERVENTIONS:
Other: Resistance Exercise — Participants will perform 4 sets of 12 repetitions of moderate intensity leg extension

SUMMARY:
Obesity has numerous comorbidities that are associated with exceedingly high healthcare costs. In addition to well- characterized impairments in lipid and glucose metabolism, obesity is associated with altered protein metabolism. We have recently observed that obese individuals are essentially nonresponsive to protein ingestion with respect to myofibrillar protein synthesis. This suggests that skeletal muscle remodeling in obese individuals is impaired possibly contributing to a poor metabolic quality of muscle. Resistance exercise is known to strongly augment muscle protein synthesis in response to protein ingestion. The purpose of this research is to determine the muscle protein synthetic response during post-exercise recovery in obese individuals. Using stable isotope methodology, we will determine the postprandial muscle protein synthetic response in 14 male and female obese adults (Age: 20-45, BMI: 30-39.9 kg/m2) immediately after an acute bout of resistance exercise. Participants will be sedentary (< 60 min exercise/ week) and weight stable for a minimum of 6 months. During the testing blood and muscle samples will be collected. In addition participants will be asked to perform moderate intensity resistance exercise. Completion of the proposed research will identify the role of resistance exercise in the maintenance of skeletal muscle tissue after the consumption of a protein-dense meal in obese people.

DETAILED DESCRIPTION:
Baseline procedures:

A parallel group design will be used for this study. Prior to the infusion trial, participants will reported to the laboratory on two separate occasions in the morning. On the first visit, we will determine participants' body weight and height as well as body composition by dual-energy X-ray absorptiometry. Finally, participants will be familiarized with unilateral leg extension and the ten repetition maximum (10RM) procedure. On a separate occasion, each subject will arrive to the lab after an overnight fast for the determination of oral glucose tolerance in response to the consumption of 75 g glucose dissolved in 500 mL of water. At the end of this visit, we will assess participant's unilateral 10RM for leg extension. In addition, participants will be instructed to refrain from vigorous physical activity and alcohol for three days prior to the tracer infusion.

Infusion protocol On the day of the infusion trial, participants will report to the laboratory at ~0700 h after a 10 h fast. An intravenous catheter will be inserted into an antecubital vein for baseline blood sample collection, after which a primed (2 μmol·kg-1), continuous infusion (0.05 μmol·kg Lean Body Mass-1·min-1) of L-[ring-13C6]phenylalanine will be initiated (t=-180 min) and maintained until the end of the trial. A second intravenous catheter placed in a contralateral dorsal hand vein will be placed in a heated blanket for repeated arterialized blood sampling. In the post-absorptive state, muscle biopsies of the vastus lateralis are to be collected at 0 min of infusion from a non-exercised control leg (CON). Subsequently, participants will perform moderate intensity unilateral leg extension exercise. Upon completion, participants will consume 170 g of lean ground pork (36 g protein). Additional muscle biopsies will be collected from both the exercised (EX) and CON legs at 120 and 300 min after pork ingestion. Arterialized blood samples will be collected every 30 or 60 min during the post-absorptive and postprandial-states and placed in pre-chilled EDTA tubes.

ELIGIBILITY:
1. Inclusion criteria

   * Healthy-weight adults: BMI 18-24.9 kg/m2
   * Obese adults: BMI 30-39.9 kg/m2
   * Aged between 20-45 years
   * Healthy
   * Sedentary
2. Exclusion criteria

   * Smoking
   * Allergies to pork consumption
   * Unusually high protein consumption
   * Vegetarians
   * Phenylketonuria (PKU)
   * Diagnosed GI tract diseases
   * Arthritic conditions
   * A history of neuromuscular problems
   * Previous participation in amino acid tracer studies
   * Predisposition to hypertrophic scarring or keloid formation
   * Individuals on any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
   * Irregular menstrual cycles during the previous year
   * Pregnancy
   * High BMI that is not representative of being obese (e.g. resistance trained individuals, football players)
   * Contraindications for exercise

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-05-01 (Actual)

PRIMARY OUTCOMES:
Myofibrillar protein synthesis | change over a 300 minute postprandial period
  Fractional synthesis rate of myofibrillar proteins

CONTACTS AND LOCATIONS:
Locations (1):
- Freer Hall, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No